CLINICAL TRIAL: NCT02077049
Title: Are Serious Games Promoting Mobility an Attractive Alternative to Conventional Self-training for Elderly People? A Randomized Controlled Trial.
Brief Title: Are Serious Games Promoting Mobility an Attractive Alternative to Conventional Self-training for Elderly People?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Klinik Valens (Other)
Collaborators: State Secretariat for Education Research and Innovation, Switzerland (Other); Office Ambient Assisted Living (Unknown)
Responsible Party: Principal Investigator, Dr. Peter Oesch, PhD PT, Klinik Valens
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KlinikenValens_Oesch_RCT-2013; EKSG 13/081/1B (Other: Cantonal Ethics Committee St.Gallen)
Record Dates: First submitted 2014-02-06; First posted 2014-03-04 (Estimated); Last update posted 2019-02-28 (Actual); Status verified 2019-02

CONDITIONS: Mobility Limitations; Geriatric Disorder
Keywords: elderly; exercise program; self-training; mobility; computer-based learning games; serious game; balance; training adherence; training compliance; Kinect ®; Fit Bit ®
MeSH Terms: conditions — Mobility Limitation | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- serious games self-training program (Experimental): Serious games are played, using Kinect® and Fit Bit®. This program is performed during the 10 days of the intervention on a self-training basis and 2 specific time-slot (2x30 min) per day are allocated for this program.
  Interventions: Device: serious games
- Conventional self-training program (Active Comparator): conventional physical exercises are performed during the 10 days of the intervention, on a self-training basis and 2 specific time-slot (2x30 min) per day are allocated for this program.
  Interventions: Other: Conventional self-training

INTERVENTIONS:
Device: serious games — Execution of computer-based games that stimulate patient's mobility. The game is displayed on a Television (TV) screen and the patient's movements are detected by the sensors of the Kinect® camera, requiring therefore no game console.
  The Fit Bit®, a mobility tracker device, is attached at the patient's belt the whole day and measure all the trips performed and stairs climbed.
  This serious games program is instructed individually by experienced physiotherapists.
  Other Names: Kinect®; Xbox®; Windows®; Fit Bit®
  Arms: serious games self-training program
Other: Conventional self-training — Participants perform conventional physical exercises that train their balance capabilities. There are instructed by experienced physiotherapists and are adapted to each patient's physical abilities. Detailed handouts are distributed to each participants.
  Other Names: gymnastic exercises; home exercises; physical exercises
  Arms: Conventional self-training program

SUMMARY:
The main objective of this study is to determine whether elderly people in rehabilitation setting show higher adherence to self-training when using computer-based-learning games (i.e. the so called serious games) than when performing conventional exercises. Secondly the study explores to which extend balance and mobility performances vary according to the mode of self-training.

The primary study hypothesis is that elderly people practice longer and more frequently with serious games than with a conventional exercise booklet. The secondary hypothesis is that patients experience a significant higher improvement in their balance capacity by using serious games compared to patients performing conventional exercises.

DETAILED DESCRIPTION:
Background:

The Swiss population, and in Europe in general, is getting older. Due to this evolving demographic trend, the need to develop specific healthcare services for this age group is becoming crucial. From the international literature, evidence-based findings have demonstrated that physical abilities of elderly people can be increased, and institutional placement and mortality can be reduced through specific inpatient rehabilitation programs (Bachmann, Finger et al. 2010).

Adults 65 years and older should carry out aerobic physical activities for at least 150 minutes of moderate intensity or for 75 minutes of high intensity in a week. Besides it is strongly recommended that senior adults perform strengthening exercises minimum twice a week and activities promoting balance minimum thrice a week (WHO 2010; NIH 2013).

In order to increase the training intensity and thus the independence in activities of daily living, older patients admitted in Kliniken Valens are instructed with a customized self-training program, in addition to the usual rehabilitation services. As for therapist-assisted sessions, this self-training program leads to significant improvement of patient's physical performance (Olney, Nymark et al. 2006) and represents therefore a proven, efficient and cost-effective intervention for inpatient settings. However, the compliance of elderly people to execute self-training exercises varies considerably. These programs are often considered as tedious and boring, and so prematurely stopped (Phillips, Schneider et al. 2004). An alternative to increase patient's motivation could be through serious games practice. Kliniken Valens has already experienced promising results with computer-based games such as the Nintendo Wii® (Schnurr and Oesch 2012).

Methods:

In this study participants are categorized in 4 strata according to their Berg Balance Score (BBS) (≤ 44 or ≥45) and their computer skills. Subsequently they are allocated randomly either in the intervention group or in the control group. In addition to the usual rehabilitation services provided in the clinic, participants of both groups are entitled to 2 additional time-slots (2 x 30 min/day) devoted to self-training and this during the 10 days of the intervention period. This protocol ensures the same conditions for each participant to perform or not self-training exercises. For safety measures, participants with a low BBS (<45) perform the program in siting, whereas those with a higher BBS (≥45) practice in standing position (in front of a bench). The time frame of the intervention phase (from t1 to t2) lasts 10 working days and starts after self-training exercises have been instructed. In other words, t1 equates to approximately day 4 after the patient's admission in the clinic and t2 is 10 working days later, i.e. approximately day 16 after admission.

Intervention group:

The participants are instructed by experienced physiotherapists on serious games with Kinect®. Additionally, participants wear the Fit Bit® (an activity tracker device) and are encouraged to walk and climb stairs instead of using the escalator. Finally participants are asked to write down in a logbook, the frequency and duration of their self-training sessions.

Control group:

As in the usual rehabilitation services, experienced physiotherapists arrange a customized self-training program, instruct the exercises and deliver a hand-out. Additionally, patients are encouraged to walk and climb stairs instead of using the escalator. Finally participants are asked to write down in a logbook, the frequency and duration of their self-training sessions.

Data collection:

Data on self-training's intensity (primary outcome) are extracted from the logbook at post-intervention (t2) i.e. after the 10 working days of the intervention phase. The Berg Balance Scale and the Falls Efficacy Scale (secondary outcomes) are completed by a blinded researcher at pre- and post-intervention (before t1 and after t2) i.e. approximately at day 1-2 after admission and day 16-17 after admission.

Data analysis:

Data are analyzed using the statistical software for social sciences (SPSS). The statistical analysis of the two groups is performed following a normal distribution of data, with an unmatched t-test. For non-normal distributions, the Mann-Whitney U test is used.

ELIGIBILITY:
Inclusion Criteria:

1. +65 years old
2. Ability to walk independently over 20meters, with or without walking aids.
3. Self-training prescribed by the doctor
4. sufficient written and spoken knowledge of German to fill out questionnaires, with or without help.
5. Informed consent

Exclusion Criteria:

1. Cognitive impairment, defined as a Mini-Mental-State Examination (MMSE) score < 26.
2. Other limiting disorders hampering the practice of computer-based games (e.g. visual impairment, numbness, vertigo)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 54 (Actual)
Dates: Start 2014-02; Primary Completion 2015-03 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Intensity of self-training | The intensity of self-training is recorded every day and thus from the begining (t1) till the end (t2) of the intervention phase ie. during 10 working days.
  Self-training intensity is defined as the frequency of training sessions (f) multiplied by the duration (T) of each training session. The training intensity (f x T) of the 10-days intervention are summated.
  These data are recorded daily in a logbook by the patient himself from t1 (which equates to approximately day 4 after admission) till the end of the intervention (t2) i.e. 10 workings days later. The logbook is then collected for data extraction at the end of the intervention (t2), which equates to approximately day 16-17 after patient's admission in the clinic.

SECONDARY OUTCOMES:
Berg Balance Scale | The test is performed at the before the start of the intervention (t1) and again at after the end of the intervention (t2) i.e. after 10 working days
  The intervention lasts 10 working days (from t1 to t2), starting from day 4 of the patient's admission in the rehabilitation center.
  The Berg Balance Scale is a clinical test for static and dynamic balance abilities. It is assessed before the start of the intervention (t1), i.e. approximately at day 1-2 after admission and again at the end of the intervention phase (t2) 10 working days later, i.e. approximately at day 16-17 after admission.
Falls Efficacy Scale - International version | The questionnaire is completed at the before the start of the intervention (t1) and again at after the end of the intervention (t2) i.e. after 10 working days
  The intervention phase lasts 10 working days (from t1 to t2), starting from day 4 of the patient's admission in the rehabilitation center.
  The Falls Efficacy Scale is a questionnaire measuring the fear of falling. It is assessed before the start of the intervention (t1), i.e. approximately at day 1-2 after admission and again at the end of the intervention phase (t2) 10 working days later, i.e. approximately at day 16-17 after admission.
Local dynamic stability | The test is performed at the before the start of the intervention (t1) and again at after the end of the intervention (t2) i.e. after 10 working days.
  Local Dynamic Stability (LDS), a non-linear gait stability index, has been advocated as an early indicator of risk for falls. LDS is measured with a tri-axial accelerometer and quantified by calculating Lyapunov exponent.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Oesch, PhD PT, Principal Investigator — Kliniken Valens
Locations (1):
- Walenstadtberg Klinik, Walenstadtberg, Canton of St. Gallen, Switzerland

REFERENCES:
- [Background] Schnurr B, & Oesch P. Sind Nintendo Wii-Balancespiele eine machbare Alternative zum herkömmlichen Selbsttraining des Gleichgewichts nach Schlaganfall? Ergoscience (4): 147-156, 2012.
- [Background] Bachmann S, Finger C, Huss A, Egger M, Stuck AE, Clough-Gorr KM. Inpatient rehabilitation specifically designed for geriatric patients: systematic review and meta-analysis of randomised controlled trials. BMJ. 2010 Apr 20;340:c1718. doi: 10.1136/bmj.c1718. PMID 20406866
- [Background] Global Recommendations on Physical Activity for Health. Geneva: World Health Organization; 2010. Available from http://www.ncbi.nlm.nih.gov/books/NBK305057/ PMID 26180873
- [Background] Phillips EM, Schneider JC, Mercer GR. Motivating elders to initiate and maintain exercise. Arch Phys Med Rehabil. 2004 Jul;85(7 Suppl 3):S52-7; quiz S58-9. doi: 10.1016/j.apmr.2004.03.012. PMID 15221728
- [Background] Olney SJ, Nymark J, Brouwer B, Culham E, Day A, Heard J, Henderson M, Parvataneni K. A randomized controlled trial of supervised versus unsupervised exercise programs for ambulatory stroke survivors. Stroke. 2006 Feb;37(2):476-81. doi: 10.1161/01.STR.0000199061.85897.b7. Epub 2006 Jan 12. PMID 16410482
- [Derived] Oesch P, Kool J, Fernandez-Luque L, Brox E, Evertsen G, Civit A, Hilfiker R, Bachmann S. Exergames versus self-regulated exercises with instruction leaflets to improve adherence during geriatric rehabilitation: a randomized controlled trial. BMC Geriatr. 2017 Mar 23;17(1):77. doi: 10.1186/s12877-017-0467-7. PMID 28330455
- [Derived] Hasselmann V, Oesch P, Fernandez-Luque L, Bachmann S. Are exergames promoting mobility an attractive alternative to conventional self-regulated exercises for elderly people in a rehabilitation setting? Study protocol of a randomized controlled trial. BMC Geriatr. 2015 Sep 7;15:108. doi: 10.1186/s12877-015-0106-0. PMID 26346751